CLINICAL TRIAL: NCT06616662
Title: Comparative Outcomes of Ligation of the Intersphincteric Fistula Tract and Mucosal Advancement Flap Techniques in Elderly Patients with Transsphincteric Perianal Fistulas: Recurrence, Incontinence and Risk Factors
Brief Title: Transsphincteric Fistula Management Using LIFT and MAF
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof of general and laparoscopic surgery, Zagazig University
Other Study IDs: perianal fistula
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Perianal Fistula
Keywords: perianal fistula,flap,ligation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LIFT
  Interventions: Procedure: LIFT
- MAF
  Interventions: Procedure: MAF

INTERVENTIONS:
Procedure: MAF — use mucosal advancement flap to treat PAF
  Groups: MAF
Procedure: LIFT — use LIFT surgery for treating PAF
  Groups: LIFT

SUMMARY:
a study that detect the most suitable surgical techniques for treating transsphincteric fistula

DETAILED DESCRIPTION:
we compared between LIFT and MAF in elderly with PAF

ELIGIBILITY:
Inclusion Criteria:

* elderly persons with PAF

Exclusion Criteria:

* recurrent fistula
* associated autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: two hundred and fifty seven elderly patient with PAF
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
healing rate | three years
  incidence of healing in both approaches

SECONDARY OUTCOMES:
incontinence | three years
  incidence of incontinence after both approaches

CONTACTS AND LOCATIONS:
Overall Officials: Tamer. A.A.M. Habeeb, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Medicine Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habeeb TAAM, Chiaretti M, Kryvoruchko IA, Pesce A, Kechagias A, Elias AA, Adam AAM, Gadallah MA, Ali Ahmed SM, Khyrallh A, Alsayed MH, Tharwat Kamel Awad E, Elshafey MH, Abo Alsaad MI, Ali AK, Elbelkasi H, Abou Zaid MA, Youssef HAA, Al-Zamek MMF, Fiad A, Elshahidy TM, Elballat MR, El Taher AK, Mohamed MMM, AboZeid AK, Mansour MI, Yassin MA, Arafa AS, Lotfy M, Mousa B, Atef B, Naguib SM, Heggy IA, Elnemr M, Zaitoun MA, AbdAllah ES, Moussa MS, Hamed AEM, Elsayed RS. Mucosal advancement flap versus ligation of the inter-sphincteric fistula tract for management of trans-sphincteric perianal fistulas in the elderly: a retrospective study. Int J Colorectal Dis. 2025 Mar 12;40(1):61. doi: 10.1007/s00384-025-04846-5. PMID 40072575